CLINICAL TRIAL: NCT07011810
Title: Axatilimab for Sclerotic Chronic Graft-Versus-Host Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125196; NCI-2025-01612 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020804 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — axatilimab; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (axatilimab) (Experimental): Patients receive axatilimab IV over 30 minutes on days 1 and 15 of cycles 1-6 and then on day 1 of remaining cycles. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection throughout the study. Additionally, patients may undergo optional skin biopsies and optional skin flexibility assessments throughout the study.
  Interventions: Biological: Axatilimab; Procedure: Biospecimen Collection; Other: Questionnaire Administration; Procedure: Skin Biopsy; Procedure: Skin Measurement

INTERVENTIONS:
Biological: Axatilimab — Given IV
  Other Names: Anti-M-CSFR Monoclonal Antibody SNDX-6352; Axatilimab-csfr; INCA 034176; INCA 34176; INCA-034176; INCA-34176; INCA034176; INCA34176; Niktimvo; SNDX 6352; SNDX-6352; SNDX6352; UCB6352
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Ancillary studies
Procedure: Skin Biopsy — Undergo optional skin biopsy
  Other Names: Biopsy of Skin
Procedure: Skin Measurement — Undergo optional skin flexibility assessment
  Other Names: Myoton PRO

SUMMARY:
This phase II trial tests how well axatilimab works in treating patients with thickening or hardening (sclerosis) of the skin related to chronic graft-versus-host disease after a donor stem cell transplant. Chronic graft-versus-host disease (cGVHD) remains a major complication of donor stem cell transplants. Sclerosis, while not associated with a higher risk of death, can lead to serious disabilities. Usual treatments for cGVHD can be associated with significant side effects and unsatisfactory outcomes. A monoclonal antibody, like axatilimab, is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Axatilimab blocks a receptor and depletes cells that may be involved in the development of inflammation and fibrosis in cGVHD. Giving axatilimab may improve or prevent worsening of sclerosis related to cGVHD in patients after a donor stem cell transplant.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive axatilimab IV over 30 minutes on days 1 and 15 of cycles 1-6 and then on day 1 of remaining cycles. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection throughout the study. Additionally, patients may undergo optional skin biopsies and optional skin flexibility assessments throughout the study.

After completion of study treatment, patients are followed up at 30 days then for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Ability to understand and willingness to sign a written informed consent document
* Allogeneic stem cell transplant, with active cGVHD requiring systemic treatment. Active cGVHD is defined as the presence of signs and symptoms of cGVHD diagnosed per the 2014 National Institutes of Health (NIH) Consensus Development Project on Criteria for Clinical trials in cGVHD
* Sclerotic skin score 2-3 or PROM < 24 due to cGVHD
* Initial diagnosis of sclerosis within the past 24 weeks (168 days)
* No new non-corticosteroid systemic immunosuppressive agent within 28 days prior to screening, unless there is a plan to stop them no later than 21 days after the first dose of axatilimab. Receipt of systemic corticosteroids ≤ 1 mg/kg prednisone or prednisone equivalent daily is allowed at the time of enrollment and may be continued after axatilimab initiation
* If patient has been previously treated with systemic immunosuppression for sclerosis, one of the following two conditions must be true: (a) the systemic immunosuppressive treatment(s) were given for at least 60 days and the sclerotic cGVHD either did not respond or progressed; (b) the systemic immunosuppressive treatment(s) were given for less than 60 days due to lack of sclerotic cGVHD response, sclerotic cGVHD progression, toxicity or logistic reasons and have or will be stopped no later than 21 days after the first dose of axatilimab
* Karnofsky performance status ≥ 60%
* Absolute neutrophil count ≥ 1.0 x 10^9/L (evaluated during the 28-day screening period)
* Platelet count ≥ 50 x 10^9/L (evaluated during the 28-day screening period) (without transfusion within 2 weeks of study entry)
* If no suspected or proven liver cGVHD, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN) (evaluated during the 28-day screening period) unless due to Gilbert's disease
* If no suspected or proven liver cGVHD, total bilirubin ≤ 1.5 x ULN (evaluated during the 28-day screening period) unless due to Gilbert's disease
* For patients with suspected or documented liver cGVHD, ALT and AST ≤ 5 x ULN (evaluated during the 28-day screening period) unless due to Gilbert's disease
* For patients with suspected or documented liver cGVHD, total bilirubin ≤ 1.5 x ULN (evaluated during the 28-day screening period) unless due to Gilbert's disease
* Estimated creatinine clearance ≥ 30 mL/min/1.73m^2 based on the institutional formula
* Male and female participants of reproductive potential must be willing to employ highly effective and acceptable forms of contraception from screening through 90 days after the last dose of study treatment.

  * Adolescent and adult male patients capable of fathering a child who are non-sterilized and who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use two methods of birth control from the time of screening throughout the total duration of the study intervention treatment period and 90 days after the last dose of study intervention. Male patients should refrain from sperm donation throughout this period
  * Female patients of childbearing potential who are not abstinent and intend to be sexually active with a non-sterilized male partner must use at least one highly effective method of contraception from the time of screening throughout the total duration of the study intervention treatment period and 90 days after the last dose of study intervention. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Female patients should also refrain from breastfeeding throughout this period
  * Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to treatment initiation. Females of childbearing potential are defined as sexually mature females without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, females who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression

Exclusion Criteria:

* Hospitalization for evaluation or management of an infection within 28 days prior to screening
* History or other evidence of significant organ dysfunction that would make the patient, in the opinion of the investigator, unsuitable for the study
* On more than 1 mg/kg/day prednisone or prednisone equivalent
* History of non-compliance
* History or other evidence of uncontrolled psychiatric illness that that would limit compliance with study requirements
* Receipt of an investigational agent within 28 days prior to screening
* Any evidence (histologic, cytogenetic, molecular, hematologic, or mixed) of relapse of the underlying cancer or post-transplant lymphoproliferative disease at the time of screening
* Diagnosed with another malignancy (other than malignancy for which transplant was performed) within 3 years of study enrollment, unless previously treated with curative intent (e.g. complete resected basal or squamous cell carcinoma of the skin)
* Active hepatitis B (defined as hepatitis B virus [HBV] surface antigen positive and HBV core antibody positive, with positive HBV deoxyribonucleic acid [DNA], or HBV positive core antibody alone with positive HBV DNA) or hepatitis C (defined as positive hepatitis C [HCV] antibody with positive HCV ribonucleic acid [RNA])
* Suspected active or latent tuberculosis (as confirmed by a positive QuantiFERON® test or other tuberculosis blood test)
* History of acute or chronic pancreatitis
* History of myositis
* Pregnant or breastfeeding
* Previous exposure to colony stimulating factor 1 receptor (CSF-1R) therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2028-08-10 (Estimated); Study Completion 2030-02-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) in sclerotic manifestations | Up to 24 weeks, cycle 7 day 1 (cycle length = 28 days)
  Will be defined as the proportion of patients with objective response per 2014 National Institutes of Health (NIH) skin and joint criteria.

SECONDARY OUTCOMES:
Failure-free survival | Up to 2 years
  Will be defined as survival free from addition of another systemic chronic graft-versus-host disease treatment, relapse or death. Kaplan Meier curves will be generated.
Modified Lee Symptom Scale summary score | Up to 2 years
  The modified Lee symptom scale will be scored according to the recommendation of the developer. A change in the summary score between baseline and follow up of ≥ 6 points will be considered clinically meaningful.
ORR in sclerotic manifestations | Up to and at cycle 13 day 1, 48 weeks (cycle length = 28 days)
  Will be defined as the proportion of patients with objective response per 2014 NIH skin and joint criteria.
Change in patient 0-10 sclerotic scale | Up to and at cycle 7 day 1 (24 weeks) and cycle 13 day 1 (48 weeks) (cycle length = 28 days)
  Will be defined as the proportion who change by 2 or more points. A change of 2 points on this scale is considered clinically meaningful.
Change in clinician 0-10 sclerotic scale | Up to and at cycle 7 day 1 (24 weeks and cycle 13 day 1 (48 weeks) (cycle length = 28 days)
  Will be defined as the proportion who change by 2 or more points. A change of 2 points on this scale is considered clinically meaningful.
ORR in all manifestations | Up to and at cycle 7 day 1 (24 weeks and cycle 13 day 1 (48 weeks) (cycle length = 28 days)
  Will be defined as the proportion of patients with objective response per 2014 NIH criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J. Lee, MD, MPH, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No